CLINICAL TRIAL: NCT04139070
Title: Electrochemotherapy for Non-curable Gastric Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REG-033-2019
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Gastric Cancer
Keywords: Electrochemotherapy; Palliative treatment
MeSH Terms: conditions — Stomach Neoplasms | interventions — Bleomycin; Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treátment group (Experimental): 8 patients are expected to be included in this study. The patients will be treated once with bleomycin in combination with elektroporation
  Interventions: Drug: Bleomycin

INTERVENTIONS:
Drug: Bleomycin — Electroporation in combination with systemically administered bleomycin
  Other Names: Electroporation

SUMMARY:
This is an explorative, phase I clinical trial. The aim of this study is to establish the safety and efficacy of electrochemotherapy for non-curable gastric cancer.

DETAILED DESCRIPTION:
This is an explorative, phase I clinical trial. Aim of this study is to establish the safety of electrochemotherapy as a palliative treatment for advanced (non-curable) gastric cancer. The study involves recruitment of 8 patients with histologically verified and non-curable gastric cancer (including Siewert Type II and II). Patients will be recruited from Department of Surgery, Odense University Hospital and from Zealand University Hospital after their case has been reviewed by the multidisciplinary team (MDT). Electrochemotherapy will take place at Department of Surgery, Zealand University Hospital. After the treatment patients will be referred to Odense University Hospital for follow-up. Electrochemotherapy will be performed as an additive treatment to standard oncological care. Patients are treated once and will be followed with endoscopy, biopsies, scans, blood samples and questionnaires after 4-6 weeks and 8-12 weeks with a minimum interval of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be mentally capable of understanding the information given.
* Patients must give written informed consent.
* Histologically verified gastric cancer (adenocarcinoma, including Siewert Type II and II)
* Non-curable disease according to MDT decision
* Age ≥ 18 years.
* ASA class I-III (Classification of the American Society of Anesthesiology)
* Thrombocytes ≥ 50 billions/l, INR >1,2. Medical correction is allowed, e.g. correction of elevated INR by means of vitamin K or administration of freshly frozen plasma.
* Performance status ECOG/WHO ≤2

Exclusion Criteria:

* Locally advanced non-metastatic EGJ/GC patients that may become resectable after pretreatment
* Inability to perform upper endoscopy with attached equipment.
* Uncorrectable coagulation disorder
* Patients with ICD or pacemaker units
* Myocardial insufficiency, defined as NYHA class >2
* Concurrent treatment with an investigational medicinal product.
* Renal impairment, defined as GFR <40 ml/min
* Pregnancy
* Concurrent inclusion in a medical trial where the intervention may affect safety measures used in the current protocol.
* Patients with any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study recruitments.
* Acute pulmonary infection.
* Medical history of severe pulmonary disease.
* Previous allergic reactions to bleomycin.
* Previous cumulative dose of bleomycin exceeding 250mg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (CTCAE) | 3 months
  Safety evaluation will be performed via continuous assessment of safety parameters by reviewing events as they arise. The investigation will be put on hold if unacceptable safety issues are outstanding.
  Adverse Events (AE) and Serious Adverse Events (SAE) will be evaluated and graded according to Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Histopathological characterization of tumor biopsies | 3 months
  Endoscopic biopsies will be collected. Standard histology (Characterization of tumor tissue, fibrosis) will be performed and regression grade according to current standards
Gene expression analysis | 3 months
  Specific immunohistochemical staining for PD-1/PD-L1, additionally, samples will be stained for CD3, CD8 and CD28. Finally, gene expression analyses will be performed using the Nano String method. In this current study, we plan to use the PanCancer IO 360 gene expression panel to analyze mRNA. This is a - 770-plex gene expression panel covering the complex interplay between tumor, microenvironment and immune response in cancer, including T and B cell activation and inhibition,, adhesion molecules, chemokines and cytokines, and pattern recognition receptors. This is a predefined gene panel and does not involve extensive mapping of the human genome.
Quality of life with "The European Organization for Research and Treatment of Cancer quality of life questionnaire" (EORTC QLQ-C30) | 3 months
  Quality of Life questionnaires will be collected at baseline and after 8-12 weeks using the EORTC QLQ-C30 questionnaire. The questionnaire consist of 30 questions with a maximum score of 126 points and a minimum score of 30 points.
Tumor volume | 3 months
  Tumor response will be evaluated through endoscopic ultrasound (EUS) to measure tumor volume before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: ismail Gögenur, DMSc, Principal Investigator — Zealand University Hospital
Locations (1):
- Department of Surgery, Zealand University Hospital, Køge, Denmark